CLINICAL TRIAL: NCT06461533
Title: General Use-results Survey of OBIZER for I.V. Injection (All-case Surveillance)
Brief Title: A Survey of Susoctocog Alfa (Genetical Recombination) in Participants With Acquired Haemophilia A
Status: Recruiting | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: TAK-672-4004
Record Dates: First submitted 2024-06-07; First posted 2024-06-17 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Acquired Hemophilia A
MeSH Terms: conditions — Factor 8 deficiency, acquired

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Susoctocog Alfa (Genetical Recombination): Participants will receive Susoctocog Alfa (Genetical Recombination) intravenous injection.
  Interventions: Drug: Susoctocog Alfa (Genetical Recombination)

INTERVENTIONS:
Drug: Susoctocog Alfa (Genetical Recombination) — Susoctocog Alfa (Genetical Recombination), Intravenous injection
  Other Names: OBIZUR Intravenous Injection 500; TAK-672

SUMMARY:
This study is a survey in Japan of Susoctocog Alfa (Genetical Recombination) intravenous injection used to treat participants with bleeding events of acquired Haemophilia A (AHA). The study sponsor will not be involved in how the participants are treated but will provide instructions on how the clinics will record what happens during the study.

The main aim of the study is to check for side effects related from Susoctocog Alfa (Genetical Recombination) intravenous injection and to check if Susoctocog Alfa (Genetical Recombination) intravenous injection improves bleeding events of AHA.

During the study, participants with AHA will take Susoctocog Alfa (Genetical Recombination) intravenous injection according to their clinic's standard practice. The study doctors will check for side effects from Susoctocog Alfa (Genetical Recombination) intravenous injection for up to 90 days after the last dose of study drug or until discontinued (varied from participant to participant).

ELIGIBILITY:
Inclusion Criteria:

- All participants with Acquired Haemophilia A, treated with Susoctocog Alfa (Genetical Recombination).

Exclusion Criteria:

- None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The population of this survey are all participants who meet the inclusion/exclusion criteria.
Sampling Method: Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2024-06-10 (Actual); Primary Completion 2029-10-31 (Estimated); Study Completion 2029-10-31 (Estimated)

PRIMARY OUTCOMES:
Number of Participants who Experience at Least One Treatment-Emergent Adverse Events (TEAE) | From first dose of study drug up to 90 days after the last dose of study drug or until discontinued, whichever came first (varied from participant to participant)
  An adverse event (AE) is defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment.
Number of Participants Who Experience at Least One Adverse Drug Reactions (ADRs) | From first dose of study drug up to 90 days after the last dose of study drug or until discontinued, whichever came first (varied from participant to participant)
  An adverse event (AE) is defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment. Adverse drug reaction refers to AE related to administered drug.

SECONDARY OUTCOMES:
Number of Participants with Each Score of Eastern Cooperative Oncology Group (ECOG) Performance Status | Pre-dose, at the last dose or discontinuation of study drug, whichever came first, and 90 days after the last dose or discontinuation of study drug, whichever came first (varied from participant to participant)
  ECOG scale will be used to assess performance status of participants. ECOG is a grade, where grade 0: Normal activity. Grade 1: Symptoms but ambulatory. Grade 2: In bed <50% of the time. Grade 3: In bed >50% of the time. Grade 4: 100% bedridden. Grade 5: Dead.
Number of Participants for Categories of Treatment Effectiveness with Susoctocog Alfa (Genetical Recombination) as Assessed by the Investigator | 24 hours after the first dose of study drug, and the last dose for bleeding episode or discontinuation of study drug, whichever came first (varied from participant to participant)
  Number of participants for categories of treatment effectiveness with Susoctocog Alfa (Genetical Recombination) will be reported. Investigator will assess participants with following categories; Effective (Bleeding stopped and Clinically controlled), Partially Effective (Blood loss decreased, and Clinically stable, improvement, or bleeding for the other reason), Ineffective (Blood loss slightly decreased or unchanged and Clinically unstable), Not Effective (Worsening of bleeding and Clinically worsening).

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- Takeda selected site, Tokyo, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/